CLINICAL TRIAL: NCT03602157
Title: Phase I Study of the Administration of T Lymphocytes Co-Expressing the CD30 Chimeric Antigen Receptor (CAR) and CCR4 for Relapsed/Refractory CD30+ Hodgkin Lymphoma and Cutaneous T-Cell Lymphoma
Brief Title: Study of CAR-T Cells Expressing CD30 and CCR4 for r/r CD30+ HL and CTCL
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Stand Up To Cancer (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1606-ATL; R01CA247497 (NIH)
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma; Immune System Diseases; Immunoproliferative Disorders; Lymphatic Diseases; Lymphoproliferative Disorders; Neoplasms; Cutaneous Lymphoma; Cutaneous Anaplastic Large Cell Lymphoma; Mycosis Fungoides; Sezary Syndrome; Lymphomatoid Papulosis; Cutaneous T Cell Lymphoma; Gray Zone Lymphoma
Keywords: CAR T cells; CD30; CCR4; Lymphoma; T lymphocytes
MeSH Terms: conditions — Lymphoma; Immune System Diseases; Immunoproliferative Disorders; Lymphatic Diseases; Lymphoproliferative Disorders; Neoplasms; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Lymphomatoid Papulosis | interventions — Bendamustine Hydrochloride; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ATLCAR.CD30.CCR4 & ATLCAR.CD30 (Experimental): A 3+3 design in adult subjects. Subjects in the first dose level will receive ATLCAR.CD30.CCR4 cells alone, once safety has been established, the initial dose of ATLCAR.CD30.CCR4 will be combined with a fixed dose of ATLCAR.CD30 cells in the next dose level. Every time the dose of ATLCAR.CD30.CCR4 is escalated, subjects in that dose level will receive ATLCAR.CD30.CCR4 alone prior to subsequent dose level enrolling subjects to receive a combination of fixed dose ATLCAR.CD30 and the selected dose level of ATLCAR.CD30.CCR4. The six dose levels will consist of: dose level 1 = 2 × 10^7 ATLCAR.CD30.CCR4 cells/m2; dose level 2 = 1 × 10^8 ATLCAR.CD30 cells/m2 and 2 × 10^7 ATLCAR.CD30.CCR4 cells/m2; dose level 3 = 5 × 10^7/m2 ATLCAR.CD30.CCR4 cells/m2; dose level 4 = 1 × 10^8 ATLCAR.CD30 cells/m2 and 5 × 10^7 ATLCAR.CD30.CCR4 cells/m2; dose level 5 = 1 × 10^8/m2 ATLCAR.CD30.CCR4 cells/m2; dose level 6 = 1 × 108 ATLCAR.CD30 cells/m2 and 1 × 108 ATLCAR.CD30.CCR4 cells/m2.
  Interventions: Biological: ATLCAR.CD30.CCR4 cells; Biological: ALTCAR.CD30 cells; Drug: Bendamustine; Drug: Fludarabine

INTERVENTIONS:
Biological: ATLCAR.CD30.CCR4 cells — Three dose levels are being evaluated: 2x10^7, 5x10^7, 1x10^8
Biological: ALTCAR.CD30 cells — Fixed dose level of 1x10^8
Drug: Bendamustine — 70 mg/m^2/day Bendamustine for 3 days for lymphodepletion prior to cell infusion
Drug: Fludarabine — 30 mg/m^2/day Fludarabine for 3 days for lymphodepletion prior to cell infusion

SUMMARY:
The body has different ways of fighting infection and disease. No single way is perfect for fighting cancer. This research study combines two different ways of fighting disease: antibodies and T cells. Antibodies are proteins that protect the body from disease caused by bacteria or toxic substances. Antibodies work by binding bacteria or substances, which stops them from growing and causing bad effects. T cells, also called T lymphocytes, are special infection-fighting blood cells that can kill other cells, including tumor cells or cells that are infected with bacteria or viruses. Both antibodies and T cells have been used to treat patients with cancers. They both have shown promise, but neither alone has been sufficient to treat cancer. This study will combine both T cells and antibodies in order to create a more effective treatment called Autologous T Lymphocyte Chimeric Antigen Receptor cells targeted against the CD30 antigen (ATLCAR.CD30). Another treatment being tested includes the Autologous T Lymphocyte Chimeric Antigen Receptor cells targeted against the CD30 antigen with CCR4 (ATLCAR.CD30.CCR4) to help the cells move to regions in the patient's body where the cancer is present. Participants in this study will receive either ATLCAR.CD30.CCR4 cells alone or will receive ATLCAR.CD30.CCR4 cells combined with ATLCAR.CD30 cells.

Previous studies have shown that a new gene can be put into T cells that will increase their ability to recognize and kill cancer cells. The new gene that is put in the T cells in this study makes an antibody called anti-CD30. This antibody sticks to lymphoma cells because of a substance on the outside of the cells called CD30. Anti-CD30 antibodies have been used to treat people with lymphoma but have not been strong enough to cure most patients. For this study, the anti-CD30 antibody has been changed so instead of floating free in the blood it is now joined to the T cells. When an antibody is joined to a T cell in this way it is called a chimeric receptor. These CD30 chimeric (combination) receptor-activated T cells (ATLCAR.CD30) can kill some of the tumor, but they do not last very long in the body and so their chances of fighting the cancer are unknown.

Researchers are working to identify ways to improve the ability of ATLCAR.CD30 to destroy tumor cells. T cells naturally produce a protein called CCR4 which functions as a navigation system directing T cells toward tumor cells specifically. In this study, researchers will also genetically modify ATLCAR.CD30 cells to produce more CCR4 proteins and they will be called ATLCAR.CD30.CCR4. The study team believes that the ATLCAR.CD30.CCR4 cells will be guided directly toward the tumor cells based on their navigation system. In addition, the study team believes the majority of ATLCAR.CD30 cells will also be guided directly toward tumor cells when given together with ATLCAR.CD30.CCR4, increasing their anti-cancer fighting ability.

This is the first time ATLCAR>CD30.CCR4 cells or combination of ATLCAR.CD30.CCR4 and ATLCAR.CD30 cells are used to treat lymphoma. The purpose of this study to determine the following:

* What is the safe dose of ATLCAR.CD30.CCR4 cells to give to patients
* What is the safe dose of the combination of ATLCAR.CD30 and ATLCAR.CD30.CCR4 cells to give to patients

DETAILED DESCRIPTION:
This study is a single center, open-label Phase I clinical trial designed to determine the safety of escalating doses of autologous activated T lymphocytes (ATLs) co-expressing the chimeric antigen receptor specific for the CD30 antigen and the CCR4 chemokine receptor (ATLCAR.CD30.CCR4) in subjects with relapsed/refractory CD30+ Hodgkin (HL) and cutaneous T Cell Lymphoma (CTCL). Subjects with grey zone lymphoma will also be eligible to enroll on this protocol; the characteristics of grey zone lymphoma are very similar to HL and therefore will be referred to collectively throughout the protocol under the general term of HL. Subjects will receive either ATLCAR.CD30.CCR4 or the ATLCAR.CD30.CCR4 product in combination with an ATL product encoding only the CAR.CD30 (ATLCAR.CD30). The dose for ATLCAR.CD30 will be fixed at the highest dose level as this product has been shown to be safe in phase I trials with and without lymphodepletion. Six total dose levels of ATLCAR.CD30.CCR4 with or without ATLCAR.CD30 will be tested. Prior to receiving the infusions, subjects will undergo lymphodepletion with bendamustine and fludarabine, The 3+3 design will be used for estimating the maximum tolerated dose (MTD) of ATLCAR.CD30.CCR4 in combination with ATLCAR.CD30. Any dose level may be expanded to 4-9 subjects to explore adverse events (AEs) of special interest prior to moving to the next dose level. If due to the expansion ≥1/3 of the total number of subject on that dose level experiences a DLT, the study would not escalate to the next highest dose level and the maximum tolerated dose would be exceeded. The final MTD will be the highest dose of ATLCAR.CD30.CCR4 and ATLCAR.CD30 with observed DLT rate of less than 1/3. An expansion cohort will enroll up to 8 subjects at the MTD of ATLCAR.CD30.CCR4 and ATLCAR.CD30 to further assess safety and efficacy of these cellular products. Secondary endpoints include evaluation of persistence of ATLCAR.CD30.CCR4 vs. ATLCAR.CD30 in the peripheral blood, accumulation of ATLCAR.CD30.CCR4 vs. ATLCAR.CD30 in tumor biopsies, and progression free survival (PFS).

LCCC1606-ATL builds on LCCC1532-ATL, a phase Ib/II trial investigating the safety and efficacy of ATLCAR.CD30 in subjects with CD30+ lymphoma.

OUTLINE

Cell Procurement

Up to 300 mL total of peripheral blood will be obtained (in up to 3 collections) from subjects for cell procurement. Up to 300 mL total of peripheral blood will be obtained (in up to 3 collections) from subjects for cell procurement. Additionally, leukapheresis may be performed to isolate sufficient cells in subjects with a low absolute lymphocyte count or who had inadequate peripheral blood collection. The parameters for apheresis will be up to 2 blood volumes. Collected peripheral blood may be used for generation of CAR-T cells if the cells were collected on another CAR-T cell trial for which Lineberger Comprehensive Cancer Center is the sponsor and if the subject is eligible for procurement/screening on the LCCC 1606-ATL protocol. ATLCAR.CD30 cells manufactured for a different protocol may be used for LCCC 1606-ATL, if they fit specifications for the protocol and the patient qualifies for the protocol.

Lymphodepletion Regimen

In order to receive lymphodepletion and CAR-T cells, subjects must still have evidence of active disease.

All subjects will receive lymphodepletion with bendamustine 70 mg/m2 and fludarabine 30 mg/m2 for 3 days to reduce possible toxicity associated with the agent prior to administration of CAR-T cells.

NOTE: Any subject who tests positive for Hepatitis B core antibody and negative for Hepatitis B viral load during screening must initiate an anti-Hepatitis B prophylaxis regimen prior to lymphodepletion.

Bendamustine and fludarabine will be administered concomitantly for lymphodepletion (i.e., intravenous (IV) administration of bendamustine 70 mg/m2/day over 3 consecutive days and IV fludarabine 30 mg/m2/day over 3 consecutive days) prior to the first CAR-T cell infusion. Bendamustine should be administered first followed by IV administration of fludarabine.

Cell Administration

ATLCAR.CD30.CCR4 with or without ATLCAR.CD30 cells will be given to eligible subjects 2-14 days (preferably 2-4 days) after lymphodepletion with fludarabine and bendamustine. The dose of cells will vary, depending on the cohort enrolled. The cells will be administered by a licensed provider (oncology nurse or physician) via intravenous injection over 1-10 minutes through either a peripheral or a central line. The expected volume will be 1-50cc. Subjects in the dose expansion part of the study who received the highest safe dose level of ATLCAR.CD30 and ATLCAR.CD30.CCR4 may receive a second infusion of ATLCAR.CD30 and ATLCAR.CD30.CCR4 if cells are available equal to the dose administered for the first cell infusion (or a lower dose).

Duration of Therapy

Therapy in LCCC1606-ATL involves one to two infusion(s) of ATLCAR.CD30.CCR4 with or without ATLCAR.CD30 cells. Treatment with one infusion will be administered unless:

* Subject decides to withdraw from study treatment, OR
* General or specific changes in the subject's condition render the subject unacceptable for further treatment in the judgment of the investigator.

Duration of Follow-up

Subjects who receive a cell infusion will be followed for up to 15 years for replication competent retrovirus (RCR) evaluation or until death, whichever occurs first. Subjects who are removed from study and do not receive the cellular therapy product due to unacceptable adverse events will be followed until resolution or stabilization of the adverse event. Subjects who have progressive disease or initiate another cancer therapy after receiving a cell infusion(s) will still be required to complete abbreviated follow up procedures.

ELIGIBILITY:
Inclusion Criteria

* Unless otherwise noted, subjects must meet all of the following criteria to participate in this study:
* Written informed consent and HIPAA authorization for release of personal health information. Subjects or their Legally Authorized Representative must sign a consent to undergo cell procurement. Written informed consent to enroll in the CAR T-cell therapy trial must be obtained prior to lymphodepletion.
* Adults ≥18 years of age.
* Subjects must have one of the following diagnoses by WHO criteria:

  * Classic Hodgkin Lymphoma
  * Mycosis fungoides
  * Sezary syndrome
  * Primary cutaneous CD30 positive T cell lymphoproliferative disorder including lymphomatoid papulosis or primary cutaneous anaplastic large cell lymphoma
  * B-cell lymphoma, unclassifiable, with features intermediate between DLBCL and classic Hodgkin Lymphoma (Grey Zone Lymphoma)
* Diagnosis of recurrent lymphoma in subjects who have failed ≥2 prior treatment regimens.
* These prior treatment regimens must include brentuximab vedotin.
* If the subject has Hodgkin Lymphoma, the subject must have either failed autologous transplant or must not be eligible for autologous transplant.
* If the subject has grey zone lymphoma, the subject must have failed an anthracycline containing regimen unless the subject was not previously a candidate for anthracycline
* Subjects relapsed after autologous or allogeneic stem cell transplant are eligible for this study.
* CD30+ disease (result can be pending at the time of cell procurement, but must be confirmed prior to treatment with ATLCAR.CD30.CCR4 and ATLCAR.CD30 cells); NOTE: CD30+ disease requires documented CD30 expression by immunohistochemistry based on the institutional hematopathology standard.
* Karnofsky score of > 60%
* For Subjects in the Expansion Cohort: Willing to undergo biopsy following the cell infusion. A biopsy may be required (i.e., considered mandatory) in subjects receiving both cellular products if the Investigator determines the tumor site is easily accessible (e.g., palpable tumor). If the Investigator feels that the biopsy would be difficult to obtain or poses a high degree of risk to the subject, it may be deferred.
* Women of childbearing potential (WOCBP) must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study, and for 6 months after the study is concluded. WOCBP are those who have not been surgically sterilized or have not been free from menses for > 1 year. The two birth control methods can be composed of: two barrier methods or a barrier method plus a hormonal method to prevent pregnancy. WOCBP subjects will also be instructed to tell their male partners to use a condom.

Exclusion Criteria

* Subjects meeting any of the following exclusion criteria will not be able to participate in this study:
* Pregnant or lactating.
* Tumor in a location where enlargement could cause airway obstruction.
* Current use of systemic corticosteroids at doses ≥10mg prednisone daily or its equivalent; those receiving <10mg daily may be enrolled at discretion of the Investigator.
* Active infection with HIV, HTLV, HCV (can be pending at the time of cell procurement; only those samples confirming lack of active infection will be used to generate transduced cells) defined as not being well controlled on therapy. Subjects are required to have negative HIV antibody, negative HTLV1 and 2 antibody, and negative HCV antibody or viral load.
* Active infection with HBV. Subjects are required to have a negative Hepatitis B surface Antigen. In addition, subjects must either have core antibody negative HBV (results can be pending at the time of cell procurement) OR if a subject is Hepatitis B core antibody positive they must have their Hepatitis B viral load checked. These subjects will be excluded if their viral load is positive at baseline. Subjects who are core antibody positive and viral load negative at baseline will be considered eligible.
* Has a known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer, or other cancer for which the subject has been disease-free for at least three years.
* A history of intolerance to fludarabine. Subjects with an intolerance to bendamustine may be allowed to enroll at the discretion of the clinical investigator if he/she thinks that the subject is a candidate for lymphodepletion with cyclophosphamide and fludarabine.
* Subject is not a good candidate for treatment with ATLCAR.CD30.CCR4 with and without ATLCAR.CD30 per Investigator's discretion.

Eligibility criteria to be met prior to procurement

Evidence of adequate organ function as defined by:

The following is required prior to procurement:

* Hgb ≥ 8.0g/dL (transfusion independent for 2 weeks prior to enrollment)
* Bilirubin ≤1.5 times the upper limit of normal (ULN). Subjects with Gilbert's syndrome may be treated despite a total bilirubin level >1.5 mg/dL if their conjugated bilirubin is <1.5× ULN
* AST ≤ 3 times ULN
* Serum creatinine ≤1.5 times ULN or Creatinine Clearance (CrCl) >60mL/min per Cockcroft and Gault
* Pulse oximetry of >90% on room air
* Imaging results from within 120 days prior to procurement to assess presence of active disease (no tumor imaging is required prior to procurement for participants with active cutaneous lymphoma).
* Negative serum pregnancy test within 72 hours prior to procurement or documentation that the subject is post-menopausal. Post-menopausal status must be confirmed with documentation of absence of menses for > 1 year, or documentation of surgical menopause involving bilateral oophorectomy.
* Subject has no clinical indication of rapidly progressing disease in opinion of treating physician.
* Subject has adequate cardiac function, defined as:

  * No ECG evidence of acute ischemia
  * No ECG evidence of active, clinically significant conduction system abnormalities
  * Prior to study entry, any ECG abnormality at screening not felt to put the subject at risk has to be documented by the Investigator as not medically significant
  * No uncontrolled angina or severe ventricular arrhythmias
  * No clinically significant pericardial disease
  * No history of myocardial infarction within the last 6 months prior to infusion
  * No Class 3 or higher New York Heart Association Congestive Heart Failure

Eligibility criteria to be met prior to lymphodepletion

* Presence of active disease. Imaging results from within 7 days prior to lymphodepletion to confirm presence of active disease. Subjects who have received bridging chemotherapy must have imaging performed at least 3 weeks after most recent therapy (imaging does not need to be repeated if it is within 7 days prior to lymphodepletion).

Evidence of adequate organ function as defined by:

The following are required prior to lymphodepletion:

* Adequate bone marrow function (ANC>1000 cells/mm3 and platelets >75,000/mm3). Subjects cannot have received platelet transfusion within 7 days of lymphodepletion.
* Bilirubin ≤1.5 times the upper limit of normal (ULN). Subjects with Gilbert's syndrome may be enrolled despite a total bilirubin level >1.5 mg/dL if their conjugated bilirubin is <1.5× ULN)
* AST ≤ 3 times ULN
* Serum creatinine ≤1.5 times ULN or Creatinine Clearance (CrCl) >60mL/min per Cockcroft and Gault
* Pulse oximetry of > 90% on room air
* Negative serum pregnancy test within 72 hours prior to lymphodepletion or documentation that the subject is post-menopausal. Post-menopausal status must be confirmed with documentation of absence of menses for > 1 year or documentation of surgical menopause involving bilateral oophorectomy.
* Subjects must have autologous transduced activated T-cells that meet the Certificate of Analysis (CofA) acceptance criteria.
* Has not received any investigational agents or received any tumor vaccines within the previous six weeks prior to lymphodepletion.
* Has not received anti-CD30 antibody-based therapy within the previous 4 weeks prior to lymphodepletion.
* Has not received chemotherapy or radiation therapy within the previous 3 weeks prior to lymphodepletion.

Subjects cannot be on strong inhibitors of CYP1A2 (e.g., fluvoxamine, ciprofloxacin) as these may increase plasma concentrations of bendamustine, and decrease plasma concentrations of its metabolites. See http://medicine.iupui.edu/clinpharm/ddis/ for an updated list of strong inhibitors of CYP1A2. (This applies to subjects who receive bendamustine for lymphodepletion (required) up through 72 hours after the last dose of bendamustine).

* Subjects who are HBV core antibody positive and HBV viral load negative prior to lymphodepletion must have initiated anti-HBV prophylaxis prior to lymphodepletion.
* Subject has no clinical indication of rapidly progressing disease in the opinion of the treating physician.
* Subject is a good candidate for treatment with ATLCAR.CD30.CCR4 with and without ATLCAR.CD30 per the investigator's discretion.

Eligibility criteria to be met prior to cell infusion after lymphodepletion

* No evidence of uncontrolled infection or sepsis.

Evidence of adequate organ function as defined by:

1. Bilirubin ≤2 times the upper limit of normal (ULN) unless attributed to Gilbert's syndrome
2. AST ≤5 times ULN
3. ALT ≤5 times ULN
4. Serum creatinine ≤3 times ULN
5. Pulse oximetry of >90% on room air

   * Subject has no clinical indication of rapidly progressing disease in the opinion of the treating physician.
   * Subject is a good candidate for treatment with ATLCAR.CD30.CCR4 with and without ATLCAR.CD30 per the investigator's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2039-11-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AE) as a measure of safety and tolerability ATLCAR.CD30.CCR4 and ATLCAR.CD30 cells | 6 weeks
  Toxicity will be classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, version 5.0), CRS toxicity will be graded according to the toxicity scale outlined in CRS Grading Criteria/Link to CRS Management Guidelines and ICANS will be graded according to the toxicity scale outlined in Management of Neurotoxicity/Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS) from CAR-T Therapy. The MTD will be based on the rate of dose-limiting toxicity.

SECONDARY OUTCOMES:
Median progression free survival (PFS) after infusion of ATLCAR.CD30.CCR4 with and without ATLCAR.CD30 in subjects with CD30+ relapsed/refractory HL and CTCL. | 15 years
  PFS is defined from day of ATLCAR.CD30.CCR4 with and without ATLCAR.CD30 infusion to relapse (in subjects in a documented complete response prior to conditioning chemotherapy) or progression (in subjects not in a complete response prior to conditioning chemotherapy), or death as a result of any cause
Median overall survival (OS) in subjects with CD30+ relapsed/refractory HL and CTCL after administration of ATLCAR.CD30.CCR4 with and without ATLCAR.CD30 | 15 years
  Overall survival will be measured from the date of administration of ATLCAR.CD30.CCR4 with and without ATLCAR.CD30 infusion to date of death
Objective response rate by 7 weeks and best overall response rate in subjects with CD30+ relapsed/refractory HL and CTCL after infusion of ATLCAR.CD30.CCR4 with and without ATLCAR.CD30 | 7 weeks
  The objective response rate will be defined as the rate of complete responses (CR) + partial responses (PR) by 7 weeks post ATLCAR.CD30.CCR4 with and without ATLCAR.CD30 infusion
The best overall response rate | 7 weeks
  The best overall response rate will be defined as the best response recorded from the start of the treatment until disease progression/recurrence or initiation of alternative therapy post ATLCAR.CD30.CCR4 with and without ATLCAR.CD30 infusion.
Differential infiltration of ATLCAR.CD30.CCR4 vs. ATLCAR.CD30 cells in tumor biopsies in subjects who received both ATLCAR.CD30.CCR4 and ATLCAR.CD30 cellular products | 15 years
  Differential infiltration of ATLCAR.CD30.CCR4 vs. ATLCAR.CD30 cells in tumor biopsies in subjects receiving both ATLCAR.CD30.CCR4 and ATLCAR.CD30 cellular products will be determined by measuring the level of the transgene and by phenotypic analyses
Persistence of ATLCAR.CD30.CCR4 vs. ATLCAR.CD30 in peripheral blood in subjects who received both ATLCAR.CD30.CCR4 and ATLCAR.CD30 cellular products | 15 years
  Persistence of ATLCAR.CD30.CCR4 and ATLCAR.CD30 cells in peripheral blood will be determined by quantitative polymerase chain reaction (PCR) and flow cytometry in samples of peripheral blood in subjects who received infusion of both ATLCAR.CD30.CCR4 and ATLCAR.CD30 cellular products

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Grover, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://unclineberger.org/